CLINICAL TRIAL: NCT00860756
Title: Sleep Disturbance in Deployed Soldiers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: LTC Mona O. Bingham, PhD, RN; Chief, Nursing Research, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: I2007.242dt
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Sleep Disturbance
Keywords: sleep; disturbance; deployment; intervention; actigraph
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Intervention Group
  Interventions: Other: Relaxation CD

INTERVENTIONS:
Other: Relaxation CD — A music CD specifically created for this study to promote effective sleep while deployed. It includes sleep instructions tailored to the military deployment environment. The CD includes a voice directed meditation component that helps focus the listener on relaxation in preparation for sleep. The second track is specifically designed music to promote slow breathing and induce sleep.

SUMMARY:
Hypotheses:

* Hypothesis 1 - Sleep can be measured in Theater using actigraph technology.
* Hypothesis 2 - Standard sleep measures in Soldiers randomized to a sleep intervention group will more closely approximate normal as compared to sleep measures of Soldiers randomized to the control group.

ELIGIBILITY:
Inclusion Criteria:

* All study participants must be on Active Duty, or be Reserve or National Guard Service Members notified of impending deployment.
* Recruited prior to deployment in order to obtain baseline measures before deployment.
* Have been stateside at least one full year.
* Able to read and speak English and consent themselves.

Exclusion Criteria:

* Subjects with self-identified sleep disorder (for example restless leg syndrome or sleep apnea)
* Pregnancy. Pregnant women will be excluded from the study since pregnancy places women in a non-deployable status and pregnant Soldiers will not be deploying.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Actigraph and self report questionnaires | baseline, 6 months, 18 months

SECONDARY OUTCOMES:
Self report questionnaires | baseline, 6 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mona O. Bingham, PhD, Principal Investigator — LTC, Chief Nursing Research Services
Locations (3):
- United States (3):
  - Evans Army Community Hospital, Fort Carson, Colorado
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas